CLINICAL TRIAL: NCT03636360
Title: The Impact of Artificial Sunlight on Human Sleep and Circadian Rhythms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Seoul Semiconductor (Unknown)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Associate Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Sunlike
Record Dates: First submitted 2018-08-02; First posted 2018-08-17 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Sleep; Circadian Dysregulation; Mood
MeSH Terms: conditions — Chronobiology Disorders | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be aware that the lighting conditions will vary during their visits, but will not be aware of the nature of the difference in the lights.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LED - Sunlike (Experimental): LED lighting with spectral pattern similar to that of sunlight
  Interventions: Device: Light
- Fluorescent (Active Comparator): Fluorescent light at same illuminance (lux) as LED light
  Interventions: Device: Light
- Dim (Placebo Comparator): Dim fluorescent light with same spectrum as "Fluorescent" condition
  Interventions: Device: Light
- LED (Active Comparator): Standard LED lighting
  Interventions: Device: Light

INTERVENTIONS:
Device: Light — 15 hours of light exposure

SUMMARY:
The purpose of this study is to examine, in healthy controls, whether LED lighting that has a color spectrum similar to that of sunlight is able to differentially impact mood, circadian rhythms, sleep, and behavior, as compared to standard fluorescent lighting.

ELIGIBILITY:
Inclusion Criteria:

* Good self-reported health
* Normal color vision

Exclusion Criteria:

* No sleep disorders
* No extreme chronotype
* Regular smoker
* Significant hearing loss
* Depression
* Alcohol use disorder
* Use of illegal drugs
* Pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Alertness | 15 hours
  Change in median reaction time score on the auditory psychomotor vigilance test
Melatonin suppression | 3 hours
  Amount of reduction in the concentration of salivary melatonin concentrations during an experimental light stimulus

SECONDARY OUTCOMES:
Mood | 15 hours
  Change in total positive and negative affect scores on the Positive and Negative Affect Schedule (PANAS)

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No